CLINICAL TRIAL: NCT01283893
Title: Standardization of D2 Lymphadenectomy and Surgical Quality Control for KLASS-02 Trial: KLASS-02-QC
Brief Title: Standardization of D2 Lymphadenectomy and Surgical Quality Control: KLASS-02-QC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2010-0637
Record Dates: First submitted 2011-01-24; First posted 2011-01-26 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Laparoscopy group: Laparoscopy group: patients who underwent laparoscopic distal gastrectomy with D2 lymphadenectomy
  Interventions: Procedure: Laparoscopic distal gastrectomy with D2 lymphadenectomy
- Open group: Open group: patients who underwent open distal gastrectomy with D2 lymphadenectomy
  Interventions: Procedure: Laparoscopic distal gastrectomy with D2 lymphadenectomy

INTERVENTIONS:
Procedure: Laparoscopic distal gastrectomy with D2 lymphadenectomy — The commonly practice laparoscopic surgery for gastric cancer involves a partial omentectomy+D1+b lymphadenectomy which includes the dissection of Lymph node stations 1, 3, 4, 5, 6, 7, 8a, 9; however, when performing a D2 lymph node dissection, a total omentectomy plus LN1, 3, 4, 5, 6, 7, 8a, 9, 12a retrieval will be completed. The same total omentectomy+D2 lymphadenectomy will also be performed by the open method.

SUMMARY:
Gastric cancer is one of the most common cancers in Korea. Having achieved excellent long-term survival for early gastric cancer patients, there is a growing interest in improving the quality of life of these patients without compromising their prognosis. Laparoscopic surgery for early gastric cancer have been found to be safe and feasible with superior short-term outcomes. Although laparoscopic gastrectomy with D2 lymphadenectomy is being performed for patients with locally advanced gastric cancer; the completeness of the D2 lymphadenectomy during laparoscopic surgery has not been evaluate and no standardized procedure exists. To conduct a clinical trial comparing laparoscopic D2 lymphadenectomy to the open approach, quality control of D2 lymphadenectomy procedure is necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have documented diagnosis of gastric cancer
* Patients receiving laparoscopic gastric cancer surgery without preoperative evidence of serosal invasion and distant lymph node metastasis as determined by evaluation of preoperative CT-scan, upper endoscopy, or endoscopic ultrasound.
* Patients undergoing gastric cancer surgery without plans for combined operations, such as resection of another organ for another primary disease.
* Patients who have received comprehensive explanation about the planned study, understand and accept all the terms of the study and willingly give consent to participate in all the required elements of the study

Exclusion Criteria:

* Patients without mental competence
* Patients who are illiterate
* Patients who are pregnant
* Patients < 20 and > 80 years old

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastric cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of operative procedure according to predetermined criteria | 6 months
  1. Video recording during the operation
  2. Peer reviewer's evaluation according to predetermined criteria
  3. Final approval by review committee
  Predetermined criteria: exact dissection of lymph node (LN) station satisfying each requirements (omentum, LN1, LN3, LN4sb, LN4d, LN5, LN6, LN7, LN8a, LN9, LN11p and LN12a)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Background] Kitano S, Shiraishi N, Fujii K, Yasuda K, Inomata M, Adachi Y. A randomized controlled trial comparing open vs laparoscopy-assisted distal gastrectomy for the treatment of early gastric cancer: an interim report. Surgery. 2002 Jan;131(1 Suppl):S306-11. doi: 10.1067/msy.2002.120115. PMID 11821829
- [Background] Kim HH, Hyung WJ, Cho GS, Kim MC, Han SU, Kim W, Ryu SW, Lee HJ, Song KY. Morbidity and mortality of laparoscopic gastrectomy versus open gastrectomy for gastric cancer: an interim report--a phase III multicenter, prospective, randomized Trial (KLASS Trial). Ann Surg. 2010 Mar;251(3):417-20. doi: 10.1097/SLA.0b013e3181cc8f6b. PMID 20160637
- [Background] Song KY, Kim SN, Park CH. Laparoscopy-assisted distal gastrectomy with D2 lymph node dissection for gastric cancer: technical and oncologic aspects. Surg Endosc. 2008 Mar;22(3):655-9. doi: 10.1007/s00464-007-9431-5. PMID 17593447
- [Background] Tokunaga M, Hiki N, Fukunaga T, Nohara K, Katayama H, Akashi Y, Ohyama S, Yamaguchi T. Laparoscopy-assisted distal gastrectomy with D2 lymph node dissection following standardization--a preliminary study. J Gastrointest Surg. 2009 Jun;13(6):1058-63. doi: 10.1007/s11605-009-0840-8. Epub 2009 Mar 7. PMID 19267164
- [Derived] Hur H, Lee HY, Lee HJ, Kim MC, Hyung WJ, Park YK, Kim W, Han SU. Efficacy of laparoscopic subtotal gastrectomy with D2 lymphadenectomy for locally advanced gastric cancer: the protocol of the KLASS-02 multicenter randomized controlled clinical trial. BMC Cancer. 2015 May 5;15:355. doi: 10.1186/s12885-015-1365-z. PMID 25939684
- [Derived] Kim HI, Hur H, Kim YN, Lee HJ, Kim MC, Han SU, Hyung WJ. Standardization of D2 lymphadenectomy and surgical quality control (KLASS-02-QC): a prospective, observational, multicenter study [NCT01283893]. BMC Cancer. 2014 Mar 19;14:209. doi: 10.1186/1471-2407-14-209. PMID 24646327